CLINICAL TRIAL: NCT01681264
Title: Effect of Guanfacine on Opioid-induced Hyperalgesia (OIH) and Tolerance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: End of NIH funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P-001510; 1R01DA036564-01 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
Keywords: Pain; Pain Management; Back pain; Neck pain
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia; Back Pain; Neck Pain | interventions — Morphine; Guanfacine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Morphine:Placebo (Active Comparator)
  Interventions: Drug: Morphine; Drug: Placebo
- Morphine:Guanfacine 1mg (Active Comparator)
  Interventions: Drug: Morphine; Drug: Guanfacine 1mg
- Morphine:Guanfacine 2mg (Active Comparator)
  Interventions: Drug: Morphine; Drug: Guanfacine 2mg
- Placebo:Guanfacine 2mg (Active Comparator)
  Interventions: Drug: Guanfacine 2mg; Drug: Placebo
- Placebo:Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine
  Other Names: MS Contin
  Arms: Morphine:Guanfacine 1mg; Morphine:Guanfacine 2mg; Morphine:Placebo
Drug: Guanfacine 1mg
  Other Names: Intuniv; Tenex
  Arms: Morphine:Guanfacine 1mg
Drug: Guanfacine 2mg
  Other Names: Intuniv; Tenex
  Arms: Morphine:Guanfacine 2mg; Placebo:Guanfacine 2mg
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Morphine:Placebo; Placebo:Guanfacine 2mg; Placebo:Placebo

SUMMARY:
Dual medication (guanfacine and morphine) as a standard treatment for chronic pain.

DETAILED DESCRIPTION:
This aim proposes that guanfacine would be a useful drug to deter Opioid-Induced Hyperalgesia (OIH) when combined with an opioid (morphine) in chronic pain management.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years old
* Chronic neck or back pain condition for at least 3 months
* VAS score of 4-8
* Has not taken an opioid for the last 3 months
* Has not taken guanfacine (or other alpha-2AR agonists) for the last 6 months

Exclusion Criteria

* Sensory deficits at site of QST, such as peripheral neuropathy
* Allergic to or has had a severe adverse reaction to study medication (i.e. opioids, guanfacine, lactose, vitamin B2 a.k.a. riboflavin)
* Cannot tolerate study drugs' maximum doses
* Takes vitamin B2 > 1.6mg/day during the study
* Pregnant or breastfeeding
* Pending litigation
* Diagnosed with Raynaud's syndrome
* Has other chronic pain conditions such as fibromyalgia or joint osteoarthritis that are predominant over back and neck pain with regard to its intensity (VAS)
* Has known pre-existing cardiovascular disease (i.e. arrhythmia - prolonged QT interval > 440ms), cerebrovascular disease, hepatic or renal impairment, CNS condition, metabolic condition, or history of syncope
* Hypotension (SBP < 90 mmHg and DBP < 60 mmHg for female or SBP < 100 mmHg and DBP < 60 mmHg for male; measured while in a sitting position) or bradycardia (resting heart rate < 60 bpm)
* Subjects are on antihypertensive drugs (e.g., a beta-blocker) that result in hypotension and/or bradycardia as defined above
* Tests positive for non-study opioids, illicit drugs, marijuana, or non-prescribed drugs
* Major psychiatric disorders that required hospitalization in the past 6 months such as: major depression, bipolar disorder, schizophrenia, anxiety disorder, or psychotic disorders
* Currently in a treatment program for alcohol or drug abuse, or currently on methadone or buprenorphine (i.e. suboxone, subutex) for treatment of addiction, or stimulants for treatment of ADHD
* History of substance or alcohol abuse (meets DSM IV criteria) per medical record or subject admission
* Subjects are on medications that serve as CYP3A4/5 inhibitors or CYP3A4 inducers including, but are not limited to, valproic acid, macrolide antibiotics, antifungal drugs, St. John wort, ACE inhibitors, nefazodone (antidepressant), calcium channel blockers, H2-receptor antagonists, anti-HIV or AIDS drugs, and antiepileptic drugs
* Subjects are on medications that are ligands for alpha2-adrenergic receptors including antipsychotic drugs (e.g. clozapine) and tricyclic or tetracyclic antidepressants (e.g. imipramine, mirtazapine, mianserin). Any medications taken by a subject at the enrollment will be reviewed regarding their compatibility with guanfacine and morphine as well as possible confounding side effects. In addition, subjects will be warned of side effects of morphine such as sedation, respiratory depression at the enrollment. Subjects will be allowed to take non-opioid pain medications except for gabapentinoids and amitriptyline/nortriptyline as far as such medications do not have incompatibility with morphine and guanfacine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | 12 weeks
  Quantitative Sensory Testing (QST) results will be used to compare the 5 treatment groups.

SECONDARY OUTCOMES:
Heat Pain Threshold | 12 weeks
  Subjects will be measured for their heat pain threshold using Quantitative Sensory Testing (QST). The testing will be done at 5 of the 6 visits.
Heat Pain Tolerance | 12 weeks
  Subjects will be measured for their heat pain tolerance using Quantitative Sensory Testing (QST). The testing will be done at 5 of the 6 visits.
Temporal Pain Summation | 12 weeks
  Subjects will be measured for their temporal pain summation using Quantitative Sensory Testing (QST). The testing will be done at 5 of the 6 visits.
Detecting Diffuse Noxious Inhibitory Control (DNIC) | 12 weeks
  Subjects will be measured for their Diffuse Noxious Inhibitory Control (DNIC). The testing will be done at 5 of the 6 visits.
Heat Sensation | 12 weeks
  Subjects will be measured for their heat sensation using Quantitative Sensory Testing (QST). The testing will be done at 5 of the 6 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Translational Pain Research, Boston, Massachusetts, United States

REFERENCES:
- See also: Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/